CLINICAL TRIAL: NCT07095517
Title: Pathways, Risk Factors, and mOleculeS to Prevent Early-onset Colorectal Tumors
Acronym: PROSPECT
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Research UK (Other)
Responsible Party: Principal Investigator, Andrew T. Chan, MD, MPH, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-460; 1OT2CA297680-01 (NIH); CGCATF-2023/100036 (Other Grant/Funding Number: Cancer Research UK)
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Cancer Prevention; Colorectal Adenoma
Keywords: colorectal cancer; colorectal cancer prevention; colorectal adenoma; obesity; incretin mimetics
MeSH Terms: conditions — Colorectal Neoplasms; Obesity | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirzepatide (Experimental): Participants will be instructed to inject tirzepatide 1 time per week for up to 24 weeks. The dose will start with a 2.5mg injection per week for the first 4 weeks. Dose will increase 2.5mg/injection every 4 weeks until 15mg/injection (or maximum tolerable dose) per week is reached.
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Study drug injected subcutaneously once a week
  Other Names: Zepbound

SUMMARY:
This research study is an open-label Phase 1 Exploratory/Pilot clinical trial to measure the effects of the incretin mimetic, tirzepatide, on tissue, urine, blood, and microbiome biomarkers associated with colorectal cancer risk and to understand the feasibility of this precision prevention trial approach for a future larger study.

DETAILED DESCRIPTION:
In this research study, we are:

* Investigating the effects of tirzepatide on biomarkers of colorectal cancer risk in patients with a recent diagnosis of adenoma, a type of intestinal polyp that can precede the development of cancer.
* Planning to measure the potential protective effects associated with tirzepatide within biological samples (biospecimens) including stool, urine, blood, and oral swab samples collected prior to, during, and after treatment with tirzepatide.
* Tirzepatide is a part of the incretin mimetic (GLP-1 receptor agonist) family, which are typically used for managing diabetes and/or obesity.
* Tirzepatide may prevent colorectal cancer through multiple possible biological mechanisms. This includes weight loss which can reduce the risk of developing obesity-associated cancers, such as colorectal cancer.
* Tirzepatide has been shown to effectively induce weight loss and improve glycemic control.

The exact mechanism by which tirzepatide acts to prevent colorectal cancer is still unknown. By performing this research study, we will study the mechanisms of its anti-cancer effect, which may lead to the discovery of novel specific characteristics (markers) that can be used to select patients for tirzepatide treatment to reduce risk of cancer in the future.

The research procedures include screening for eligibility and study treatment and scheduling four clinical research visits:

* Initial visit - immediately before starting the study drug
* Week 1 visit
* Midpoint visit (9-12 weeks later) (Midpoint visit)
* Final visit (after completing the drug intervention)

At the Initial and Final visits, a flexible sigmoidoscopy will be performed along with the collection of body measurements, questionnaire data, blood, urine, saliva, stool, and up to 24 tissue biopsy samples. The first dose of the study drug will be administered by study staff at the initial visit. Participants will self-administer the second dose of the study drug at the Week 1 visit under supervision of study staff. At the Week 1 and Midpoint visits, they will also provide body measurements, blood, urine, saliva, and stool samples.

Participants will be instructed to inject tirzepatide 1 time per week for up to 24 weeks. The dose will start with a 2.5mg injection per week for the first 4 weeks. Dose will increase 2.5mg/injection every 4 weeks until 15mg/injection (or maximum tolerable dose) per week is reached. Participants will be followed weekly during this time. In the very rare occasion that there are unavoidable issues scheduling the final visit, treatment may be extended up to an additional 4 weeks.

It is expected that about 20 people will take part in this research study.

This research is being supported by The Cancer Grand Challenges partnership funded by Cancer Research UK, the National Cancer Institute, the Bowelbabe Fund for Cancer Research UK and Institut National Du Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years Because no dosing or adverse event data are currently available on the use of tirzepatide in participants <18 years of age, children are excluded from this study. Because we are specifically studying the prevention of EOCRC, which is defined as CRC occurring prior to age 50, the study population will only enroll participants under the age of 50 at baseline.
* BMI between 27 and 40 kg/m2
* Underwent a screening or surveillance colonoscopy within the prior 9 months.
* Removal of multiple (at least 2) colon or rectal adenomas (including sessile serrated adenomas but excluding hyperplastic polyps) or a single adenoma ≥6mm in size during the last colonoscopy
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have ever taken incretin mimetic therapies.
* Participants with a history of medullary thyroid cancer or MEN 2 syndrome.
* Participants at high risk of pancreatitis or otherwise contraindicated for use of tirzepatide according to clinical labeling.
* Participants with a history of cancer (excluding non-melanoma skin) within the last three years
* Participants with a history of diabetes mellitus
* Participants with a history of bowel surgery
* Participants with hereditary cancer syndromes, including HNPCC/Lynch syndrome or familial adenomatous polyposis
* Participants with a history of inflammatory bowel disease, Crohn's, or colitis.
* Participants with incomplete or partial polypectomy during prior colonoscopy.
* Participants who are pregnant. Participants who may become pregnant or partners of those who may become pregnant while on study will receive contraception counseling. Participants or partners of those who become pregnant while participating on the study should immediately inform their doctor.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Urinary PGE-M | From enrollment to the end of treatment at 24 weeks
  To determine the effect of tirzepatide intervention on urinary prostaglandin metabolites (PGE-M), an established CRC risk biomarker, in context of changes in body weight.

SECONDARY OUTCOMES:
Change in Plasma GDF-15 | From enrollment to the end of treatment at 24 weeks
  Comparing change in GDF-15 in pre- and post-treatment plasma

OTHER OUTCOMES:
Change in Microbiome | From enrollment to the end of treatment at 24 weeks
  Comparing change in gut microbiome features (species - to strain level specificity; metabolic pathways; enzymes) and metabolites using deep meta'omic profiling in pre- and post- treatment samples.
Change in ISC Marker Gene Expression | From enrollment to the end of treatment at 24 weeks
  Assess the difference in the change of ISC marker using scRNA-seq data anlysis

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T. Chan, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: Andrew T. Chan, MD, MPH. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the MGB Innovation at PHSINNOVATIONSUPPORT@partners.org